CLINICAL TRIAL: NCT00362960
Title: Effect of Different Doses of Olmesartan Medoxomil Compared to Losartan on Proteinuria, Renal Function and Inflammatory Markers in Type 2 Diabetics With Nephropathy
Brief Title: Olmesartan Medoxomil and Diabetic Nephropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sankyo Pharma Gmbh (Industry)
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SE-866/29
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2006-10-09 (Estimated); Status verified 2006-08

CONDITIONS: Type 2 Diabetes Mellitus; Diabetic Nephropathy; Proteinuria; Renal Disease
Keywords: Type 2 Diabetes Mellitus; Diabetic Nephropathy; Inflammatory Markers; Proteinuria; Renal Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Proteinuria; Kidney Diseases | interventions — Olmesartan Medoxomil; Losartan

INTERVENTIONS:
Drug: Olmesartan medoxomil
Drug: Losartan

SUMMARY:
Evaluation of several olmesartan dosages compared to losartan on proteinuria, renal function and inflammatory markers in patients with diabetic nephropathy

ELIGIBILITY:
Inclusion Criteria:

* Male or female European out-patients
* Greater than or equal to 30 years of age
* Type 2 diabetes first diagnosed at greater than or equal to 30 years of age
* Urinary protein excretion between 200-4000 mg/day exclusive
* Mean sitting dBP less than or equal to 110 mgHg
* Medically justifiable to withdraw antihypertensive treatment due to poor tolerability or inefficacy of previous treatment, or verification that treatment is still necessary

Exclusion Criteria:

* Females pregnant, nursing or planning to become pregnant or were of childbearing potential and not using acceptable methods of contraception
* Secondary forms of hypertension other than diabetic nephropathy, malignant hypertension or patients with sitting dBP exceeding 110 mmHg or sitting sBP exceeding 200 mmHg
* ECG evidence of 2nd or 3rd degree AV-block, atrial fibrillation, cardiac arrhythmia (requiring therapy) or bradycardia
* Presence of significant cardiovascular disease
* Significant cerebrovascular disease, gastrointestinal, haematological or hepatic disease or myocardial infarction in last 12 months or a previous history of any serious underlying disease
* Concurrent renal disease, nephrectomy and/or renal transplant, serum creatinine level greater than or equal to 2.0 mg/dL or creatinine clearance CLCR less than or equal to 50 mL/min
* Clinically significant lab abnormalities (ASAT/SGOT, ALAT/SGPT and γ-GT )
* Serum potassium level < 2.5 mmol/L or > 5.5 mmol/L
* Treatment of concurrent indications with drugs or medication which could have influenced BP
* History of hypersensitivity, lack of response or contraindication to Ang II-antagonists, HCTZ or atenolol, or hypersensitivity to related drugs (cross-allergy)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2003-05; Study Completion 2004-09

PRIMARY OUTCOMES:
Efficacy of olmesartan medoxomil doses compared to losartan in
patients with type 2 diabetes and nephropathy in terms of the change in
proteinuria (total urinary protein excretion) from baseline.

SECONDARY OUTCOMES:
Efficacy of the treatment with olmesartan medoxomil dosages compared to
losartan in patients with type 2 diabetes and nephropathy in terms of
change in:
creatinine clearance (CLCR)
the protein pattern (nephelometry)
inflammatory markers (circulating serum markers).
Evaluate safety and tolerability of all treatments.

CONTACTS AND LOCATIONS:
Overall Officials: H Haller, MD, Principal Investigator — Hannover Medical School
Locations (27):
- Czechia (3):
  - Frýdlant
  - Liberec
  - Prague
- Tartu, Estonia
- Germany (3):
  - Augsburg
  - Greifenstein-Beilstein
  - Hanover
- Zwijndrecht, Netherlands
- Poland (10):
  - Grodzisk Mazowiecki
  - Krakow
  - Poznan
  - Pruszków
  - Płock
  - Torun
  - Warsaw
  - Watlack
  - Wołomin
  - Wroclaw
- Slovakia (7):
  - Banská Bystrica
  - Košice
  - Lučenec
  - Martin
  - Nitra
  - Nové Zámky
  - Šahy
- Spain (2):
  - Barcelona
  - Madrid